CLINICAL TRIAL: NCT06283940
Title: Effect of Physiotherapist-led Exercise-based Cardiac Rehabilitation in Older Patients With Aortic Stenosis Who Have Undergone TAVI?
Brief Title: Exercise-based Cardiac Rehabilitation in Patients With Aortic Stenosis After Transcatheter Aortic Valve Implantation
Acronym: TAVI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 281694
Record Dates: First submitted 2024-02-06; First posted 2024-02-28 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic valve disease; Physiotherapy; Exercise; Frailty; Quality of life
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Disease; Motor Activity; Frailty

STUDY DESIGN:
Intervention Model Description: Intervention group and matched controls based on age, gender and exercise capacity in watt.
Masking Description: Data collection will be conducted by a physiotherapist not involved in the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapist-led exercise based cardiac rehabilitation (PT-X) (Experimental): PT-X consists of centralcirculatory aerobic exercise and muscular endurance training in an existing PT-X group at Alingsas Hospital in Sweden. The patients will follow an individually tailored exercise program, twice a week for 60 minutes each session over 12 weeks. The physiotherapist guides and progresses the program based on the patient's exercise capacity throughout the intervention. Additionally, two sessions of home-based exercise will be added and recorded in an exercise diary. The exercise programs are prescribed after the patient's individual exercise capacity, with perceived exertion graded 13-17 on Borg's 6-20 scale.
  Interventions: Other: Physiotherapist-led exercise based cardiac rehabilitation (PT-X)
- Control group (No Intervention): The patient will continue with their usual activities during the control period

INTERVENTIONS:
Other: Physiotherapist-led exercise based cardiac rehabilitation (PT-X) — Individually prescribed centralcirculatory aerobic exercise and muscular endurance training twice a week for 60 minutes each session over 12 weeks in a hospital-based setting, and two sessions of home-based exercise recorded in an exercise diary.
  Arms: Physiotherapist-led exercise based cardiac rehabilitation (PT-X)

SUMMARY:
Aortic valve stenosis (AS) is the most common valve disease among older individuals. In symptomatic AS, mortality is high, and the only treatment that improves prognosis and survival is transcatheter aortic valve implantation (TAVI). TAVI is a growing treatment in Sweden, allowing previously inoperable older patients with AS, who are often frail and have comorbidities, to receive intervention. This results in the need for postoperative cardiac rehabilitation for patients treated with TAVI. Previous systematic reviews and meta-analyses examining the effect of physiotherapist-led exercise-based cardiac rehabilitation (PT-X) after TAVI have shown that participation in PT-X can improve physical fitness (the highest measured oxygen uptake (VO2peak)), walking distance, walking speed, and health-related quality of life (HR-QoL). However, the included studies are limited, and there is selection bias, resulting in low evidence. Therefore, access to PT-X is currently almost non-existent in Sweden. As more patients undergo TAVI, it is crucial to investigate whether PT-X after TAVI can further improve physical fitness, HR-QoL, and reduce hospital admissions in older individuals with AS.

Objective: Primary, to investigate whether participation in PT-X after TAVI can impact physical fitness, physical activity level, and health-related quality of life. Secondary, to study the prevalence of frailty and the number of hospital admissions during the first postoperative year after TAVI.

Expected outcome: If patients with AS who have undergone TAVI can improve physical fitness, it could potentially strengthen the evidence and optimize the patient's physical capabilities. Increased access to PT-X and awareness of frailty in these patients could reduce the risk of falls and possibly the number of hospital readmissions. This would decrease healthcare consumption and improve the patient's quality of life.

DETAILED DESCRIPTION:
Aortic valve stenosis (AS) is the most common valve disease with the highest prevalence in older individuals. Healthcare is unequal, with women receiving specialist care and interventions less frequently than men. They also receive the diagnosis later, and mortality rates are higher. AS develops over time, and in the presence of symptomatic AS such as angina pectoris, syncope, and heart failure, the prognosis is poor, and mortality is high. If untreated, AS is a disease with a 2-year relative mortality risk of 50%. In older patients at high risk with symptomatic AS, transcatheter aortic valve implantation (TAVI) is the only medical treatment that improves prognosis and survival.

Since 2008, TAVI has been performed in Sweden as a standard treatment with priority 3 in the the recommendations given by the National Board of Health and Welfare in Sweden. The number of TAVI procedures in Sweden is steadily increasing and now exceeds isolated open aortic valve surgery. This development allows patients with severe symptoms and high risk, who were previously inoperable, to undergo valve intervention.

Frailty is a condition where at least three of the following criteria should be met: involuntary weight loss, self-reported fatigue, sarcopenia, reduced physical capacity, slow walking speed, and low physical activity level. Studies show that 50-70% of those undergoing TAVI due to AS are defined as frail elderly individuals with comorbidities such as heart failure and renal failure. Furthermore, studies have demonstrated an increased risk of falls and difficulty participating in daily activities due to reduced peak oxygen uptake (VO2peak), short walking distance, lower walking speed, and impaired Health Related Quality of Life (HR-QoL). It is well-established that a low VO2peak correlates with increased risk of premature death in both healthy individuals and those with chronic disease (19). Moreover, there is a strong correlation between a short walking distance and prognosis in patients with chronic diseases.

Since patients with AS already have reduced physical fitness preoperatively, a prolonged recovery time is usually observed postoperatively. Systematic reviews and meta-analyses examining the effect of physiotherapist-led exercise-based cardiac rehabilitation (PT-X) after TAVI have shown that participation in PT-X can improve VO2peak, walking distance, walking speed, and HR-QoL. However, the included studies are few and exhibit varying study quality, leading to selection bias. Despite this, the opportunity to participate in PT-X after TAVI is virtually non-existent in Sweden due to low evidence, and national and international cardiac care guidelines do not mention the possibility of PT-X after TAVI.

This has resulted in patients who have undergone TAVI not being recommended PT-X as part of their medical treatment, unlike conditions such as heart failure and ischemic heart disease, which have high priority and high evidence. As more patients undergo TAVI, it is of utmost importance to investigate whether PT-X after TAVI can further improve physical capacity, quality of life, and reduce hospital admissions.

Objective: Primary, to investigate whether participation in PT-X after TAVI can impact physical fitness, physical activity level, and health-related quality of life. Secondary, to study the prevalence of frailty and the number of hospital admissions during the first postoperative year after TAVI.

How will participation in PT-X impact exercise capacity compared to the control group that is allowed to continue with their usual life? How will participation in PT-X impact the muscle function compared to the control group that is allowed to continue with their usual life? How will participation in PT-X impact the patients physical activity level compared to the control group that is allowed to continue with their usual life? How will participation in PT-X impact HR-QoL compared to the control group that is allowed to continue with their usual life?

Secondary Research Questions:

What is the prevalence of frailty in the study population that has undergone 12 weeks of PT-X compared to the control group? What is the incidence of hospital admissions in patients who have undergone 12 weeks of PT-X compared to the control group?

Method:

Study Population: Patients, 65 years or older, with AS who have undergone TAVI and are being followed-up at SV Alingsas Hospital will be invited to participate in an intervention study. The control group consists of matched controls based on age, gender, and exercise capacity in watts, followed up at Sahlgrenska University hospital in Gothenburg. Patients in the control group will be approached for participation by a research nurse from Sahlgrenska Universityhospital. All patients will be informed verbally and in writing, and informed consent will be obtained. The study follows the Helsinki Declaration,

Data Analysis and statistical power:

Ratio and interval data will be presented as mean ± 1 standard deviation, ordinal data as median and interquartile range, and nominal data in absolute and relative numbers.

Depending on normal distribution, Student's T-test or Mann-Whitney's U-test will be used to examine differences between groups.

Paired T-test or Wilcoxon signed-rank test will highlight within-group differences, and Chi-square test will study differences in nominal data.

Multiple regression will be used to study the relationship between group membership and the primary outcome measure, work capacity in watts.

Statistical power was calculated with an 80% power (β) to detect a statistically significant difference (α) at 5%. For the training group to achieve a significant (p=0.05) improvement of 10 watts in work capacity compared to the control group, 56 individuals must be included in each group. Considering a potential dropout of approximately 20%, a total of 135 individuals will be included in the study.

Expected Result / Clinical Significance:

If patients with AS who have undergone TAVI can improve physical fitness, it could potentially strengthen the evidence and optimize the patient's physical fitness.

Increased access to PT-X and awareness of frailty in these patients could reduce the risk of falls and possibly the number of hospital readmissions, leading to reduced healthcare consumption and increased quality of life for the patient.

Gender Perspective of the Project:

The study will include both men and women to achieve groups as similar as possible regarding gender, age, and exercise capacity in watts.

ELIGIBILITY:
Inclusion Criteria:

* Aortic stenosis treated with TAVI.

Exclusion Criteria:

* Patients who, due to another disability, cannot perform the study protocol for physical fitness, PT-X, or complete the questionnaires included in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity in watt | Baseline, after 12 weeks
  Exercise capacity will be measured by a symptom-limited ergometer cycle test based on World Health Organization (WHO) protocol, monitored with electrocardiogram (ECG), bloodpressure and heartrate.
Rating of perceived exertion Borg RPE scale 6-20 | Baseline, after 12 weeks
  Borg's Rating of Perceived Exertion (RPE scale 6-20) are recorded. The cycle test concludes when the person reaches an exertion level of 17 on Borg's scale.
Exercise capacity in Watt | 12 months after the intervention completion.
  Exercise capacity will be measured by a symptom-limited ergometer cycle test based on World Health Organization (WHO) protocol, monitored with electrocardiogram (ECG), bloodpressure and heartrate.
Rating of perceived exertion Borg RPE scale 6-20 | 12 months after the intervention completion.
  Borg's Rating of Perceived Exertion (RPE scale 6-20) are recorded. The cycle test concludes when the person reaches an exertion level of 17 on Borg's scale.
Muscular endurance test, shoulder flexion | Baseline, after 12 weeks
  A unilateral isoinertial shoulder flexion test assessed with the patient sitting on a stool with their back touching the wall holding a dumbbell in their hand, 2 kg for women and 3 kg for men. The tested arm is elevated to 90º flexion and the arm not tested is placed in the patient's knee. A pace of 40 beats per min is kept by a digital metronome.
Muscular endurance test, shoulder flexion | 12 months after the intervention completion.
  A unilateral isoinertial shoulder flexion test assessed with the patient sitting on a stool with their back touching the wall holding a dumbbell in their hand, 2 kg for women and 3 kg for men. The tested arm is elevated to 90º flexion and the arm not tested is placed in the patient's knee. A pace of 40 beats per min is kept by a digital metronome.
Muscle endurance test, shoulder abduction | Baseline, after 12 weeks
  Bilateral isometric shoulder abduction is assessed with the patient holding a 1 kg dumbbell in each hand using the same body position as above. The patient is asked to elevate both arms to 90°of shoulder abduction and to maintain this position as long as possible (measured in s).
Muscle endurance test, shoulder abduction | 12 months after the intervention completion.
  Bilateral isometric shoulder abduction is assessed with the patient holding a 1 kg dumbbell in each hand using the same body position as above. The patient is asked to elevate both arms to 90°of shoulder abduction and to maintain this position as long as possible (measured in s).
Muscle endurance test, unilateral heel-lift | Baseline, after 12 weeks
  Unilateral isoinertial heel-lift is assessed with the patients performing as many unilateral heel-lifts as possible, with a straight knee, on a 10° tilted wedge, with shoes on. A pace of 60 beats per minutes is kept is kept by a metronome.
Muscle endurance test, unilateral heel-lift | 12 months after the intervention completion.
  Unilateral isoinertial heel-lift is assessed with the patients performing as many unilateral heel-lifts as possible, with a straight knee, on a 10° tilted wedge, with shoes on. A pace of 60 beats per minutes is kept is kept by a metronome.
Lower extremity function | Baseline, after 12 weeks
  Swedish version of Short Physical Performance Battery (SPPB-S) is used to measure lower extremity function in older individuals. The scale consists of three domains, maximal points 12, lower scores indicates greater limitations.
Lower extremity function | 12 months after the intervention completion.
  Swedish version of Short Physical Performance Battery (SPPB-S) is used to measure lower extremity function in older individuals.The scale consists of three domains, maximal points 12, lower scores indicates greater limitations.
Physical activity | Baseline, after 12 weeks
  Measured using an accelerometer (Actigraph® GT3x+, Actigraph, Pensacola, Florida, USA) placed on the right hip, worn continuously for seven consecutive days, excluding showering or swimming.
Physical activity | 12 months after the intervention completion.
  Measured using an accelerometer with Actigraph® GT3x+ accelerometer placed on the right hip, worn continuously for seven consecutive days, excluding showering or swimming.
Self-assessed level of physical activity | Baseline, after 12 weeks
  Self-assessed level of physical activity is measured using the short form International Physical Activity Questionnaire (IPAQ).
Self-assessed level of physical activity | 12 months after the intervention completion.
  Self-assessed level of physical activity is measured using the short form International Physical Activity Questionnaire (IPAQ).
Health Related Quality of Life | Baseline, after 12 weeks
  Swedish version of RAND 36 is employed to measure health-related quality of life.The scale consists of eight subscales. Subscale scores ranges from 0-100, higher value represent better health status.
Health Related Quality of Life | 12 months after the intervention completion.
  Swedish version of RAND 36 is employed to measure health-related quality of life.The scale consists of eight subscales. Subscale scores ranges from 0-100, higher value represent better health status.

SECONDARY OUTCOMES:
Frailty | Baseline, after 12 weeks
  Frailty is evaluated using the Swedish version of Clinical Frailty Scale.
Frailty | 12 months after the intervention completion.
  Frailty is evaluated using the Swedish version of Clinical Frailty Scale.
Hospital admission | Baseline, after 12 weeks
  Information about the number of hospital admissions after surgery will be obtained from respective hospitals.
Hospital admission | 12 months after the intervention completion.
  Information about the number of hospital admissions after surgery will be obtained from respective hospitals.

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Borland, PhD RPT, Principal Investigator — SV Hospital group Alingsås hospital, Alingsås, Sweden
Locations (1):
- SV Hospital group Alingsås hospital, Alingsås, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vahanian A, Beyersdorf F, Praz F, Milojevic M, Baldus S, Bauersachs J, Capodanno D, Conradi L, De Bonis M, De Paulis R, Delgado V, Freemantle N, Gilard M, Haugaa KH, Jeppsson A, Juni P, Pierard L, Prendergast BD, Sadaba JR, Tribouilloy C, Wojakowski W; ESC/EACTS Scientific Document Group. 2021 ESC/EACTS Guidelines for the management of valvular heart disease: Developed by the Task Force for the management of valvular heart disease of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). Rev Esp Cardiol (Engl Ed). 2022 Jun;75(6):524. doi: 10.1016/j.rec.2022.05.006. No abstract available. English, Spanish. PMID 35636831
- [Background] Carabello BA, Paulus WJ. Aortic stenosis. Lancet. 2009 Mar 14;373(9667):956-66. doi: 10.1016/S0140-6736(09)60211-7. Epub 2009 Feb 21. PMID 19232707
- [Background] Coffey S, Roberts-Thomson R, Brown A, Carapetis J, Chen M, Enriquez-Sarano M, Zuhlke L, Prendergast BD. Global epidemiology of valvular heart disease. Nat Rev Cardiol. 2021 Dec;18(12):853-864. doi: 10.1038/s41569-021-00570-z. Epub 2021 Jun 25. PMID 34172950
- [Background] Makkar RR, Fontana GP, Jilaihawi H, Kapadia S, Pichard AD, Douglas PS, Thourani VH, Babaliaros VC, Webb JG, Herrmann HC, Bavaria JE, Kodali S, Brown DL, Bowers B, Dewey TM, Svensson LG, Tuzcu M, Moses JW, Williams MR, Siegel RJ, Akin JJ, Anderson WN, Pocock S, Smith CR, Leon MB; PARTNER Trial Investigators. Transcatheter aortic-valve replacement for inoperable severe aortic stenosis. N Engl J Med. 2012 May 3;366(18):1696-704. doi: 10.1056/NEJMoa1202277. Epub 2012 Mar 26. PMID 22443478
- [Background] Kodali SK, Williams MR, Smith CR, Svensson LG, Webb JG, Makkar RR, Fontana GP, Dewey TM, Thourani VH, Pichard AD, Fischbein M, Szeto WY, Lim S, Greason KL, Teirstein PS, Malaisrie SC, Douglas PS, Hahn RT, Whisenant B, Zajarias A, Wang D, Akin JJ, Anderson WN, Leon MB; PARTNER Trial Investigators. Two-year outcomes after transcatheter or surgical aortic-valve replacement. N Engl J Med. 2012 May 3;366(18):1686-95. doi: 10.1056/NEJMoa1200384. Epub 2012 Mar 26. PMID 22443479
- [Background] Lindman BR, Sukul D, Dweck MR, Madhavan MV, Arsenault BJ, Coylewright M, Merryman WD, Newby DE, Lewis J, Harrell FE Jr, Mack MJ, Leon MB, Otto CM, Pibarot P. Evaluating Medical Therapy for Calcific Aortic Stenosis: JACC State-of-the-Art Review. J Am Coll Cardiol. 2021 Dec 7;78(23):2354-2376. doi: 10.1016/j.jacc.2021.09.1367. PMID 34857095
- [Background] Mack MJ, Leon MB, Smith CR, Miller DC, Moses JW, Tuzcu EM, Webb JG, Douglas PS, Anderson WN, Blackstone EH, Kodali SK, Makkar RR, Fontana GP, Kapadia S, Bavaria J, Hahn RT, Thourani VH, Babaliaros V, Pichard A, Herrmann HC, Brown DL, Williams M, Akin J, Davidson MJ, Svensson LG; PARTNER 1 trial investigators. 5-year outcomes of transcatheter aortic valve replacement or surgical aortic valve replacement for high surgical risk patients with aortic stenosis (PARTNER 1): a randomised controlled trial. Lancet. 2015 Jun 20;385(9986):2477-84. doi: 10.1016/S0140-6736(15)60308-7. Epub 2015 Mar 15. PMID 25788234
- [Background] Otto CM, Prendergast B. Aortic-valve stenosis--from patients at risk to severe valve obstruction. N Engl J Med. 2014 Aug 21;371(8):744-56. doi: 10.1056/NEJMra1313875. No abstract available. PMID 25140960
- [Background] Harnek J, Nilsson J, Friberg O, James S, Lagerqvist B, Hambraeus K, Cider A, Svennberg L, Attebring MF, Held C, Johansson P, Jernberg T. The 2011 outcome from the Swedish Health Care Registry on Heart Disease (SWEDEHEART). Scand Cardiovasc J. 2013 Jun;47 Suppl 62:1-10. doi: 10.3109/14017431.2013.780389. PMID 23941732
- [Background] Cribier AG. The Odyssey of TAVR from concept to clinical reality. Tex Heart Inst J. 2014 Apr 1;41(2):125-30. doi: 10.14503/THIJ-14-4137. eCollection 2014 Apr. No abstract available. PMID 24808769
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Mack M. Frailty and aortic valve disease. J Thorac Cardiovasc Surg. 2013 Mar;145(3 Suppl):S7-10. doi: 10.1016/j.jtcvs.2012.11.063. Epub 2012 Dec 20. PMID 23260463
- [Background] Goel K, Holmes DR Jr. Transcatheter Aortic Valve Replacement: OPTIMIZING OUTCOMES FOR HEALTHY RECOVERY. J Cardiopulm Rehabil Prev. 2018 Jan;38(1):1-7. doi: 10.1097/HCR.0000000000000301. PMID 29251657
- [Background] Iung B, Delgado V, Rosenhek R, Price S, Prendergast B, Wendler O, De Bonis M, Tribouilloy C, Evangelista A, Bogachev-Prokophiev A, Apor A, Ince H, Laroche C, Popescu BA, Pierard L, Haude M, Hindricks G, Ruschitzka F, Windecker S, Bax JJ, Maggioni A, Vahanian A; EORP VHD II Investigators. Contemporary Presentation and Management of Valvular Heart Disease: The EURObservational Research Programme Valvular Heart Disease II Survey. Circulation. 2019 Oct;140(14):1156-1169. doi: 10.1161/CIRCULATIONAHA.119.041080. Epub 2019 Sep 12. PMID 31510787
- [Background] Russo N, Compostella L, Tarantini G, Setzu T, Napodano M, Bottio T, D'Onofrio A, Isabella G, Gerosa G, Iliceto S, Bellotto F. Cardiac rehabilitation after transcatheter versus surgical prosthetic valve implantation for aortic stenosis in the elderly. Eur J Prev Cardiol. 2014 Nov;21(11):1341-8. doi: 10.1177/2047487313494029. Epub 2013 Jun 11. PMID 23757283
- [Background] Izquierdo M, Merchant RA, Morley JE, Anker SD, Aprahamian I, Arai H, Aubertin-Leheudre M, Bernabei R, Cadore EL, Cesari M, Chen LK, de Souto Barreto P, Duque G, Ferrucci L, Fielding RA, Garcia-Hermoso A, Gutierrez-Robledo LM, Harridge SDR, Kirk B, Kritchevsky S, Landi F, Lazarus N, Martin FC, Marzetti E, Pahor M, Ramirez-Velez R, Rodriguez-Manas L, Rolland Y, Ruiz JG, Theou O, Villareal DT, Waters DL, Won Won C, Woo J, Vellas B, Fiatarone Singh M. International Exercise Recommendations in Older Adults (ICFSR): Expert Consensus Guidelines. J Nutr Health Aging. 2021;25(7):824-853. doi: 10.1007/s12603-021-1665-8. PMID 34409961
- [Background] Lee DC, Sui X, Artero EG, Lee IM, Church TS, McAuley PA, Stanford FC, Kohl HW 3rd, Blair SN. Long-term effects of changes in cardiorespiratory fitness and body mass index on all-cause and cardiovascular disease mortality in men: the Aerobics Center Longitudinal Study. Circulation. 2011 Dec 6;124(23):2483-90. doi: 10.1161/CIRCULATIONAHA.111.038422. PMID 22144631
- [Background] Bohannon RW, Crouch R. Minimal clinically important difference for change in 6-minute walk test distance of adults with pathology: a systematic review. J Eval Clin Pract. 2017 Apr;23(2):377-381. doi: 10.1111/jep.12629. Epub 2016 Sep 4. PMID 27592691
- [Background] Tarro Genta F. Cardiac Rehabilitation for Transcatheter Aortic Valve Replacement. Clin Geriatr Med. 2019 Nov;35(4):539-548. doi: 10.1016/j.cger.2019.07.007. Epub 2019 Jul 3. PMID 31543184
- [Background] Anayo L, Rogers P, Long L, Dalby M, Taylor R. Exercise-based cardiac rehabilitation for patients following open surgical aortic valve replacement and transcatheter aortic valve implant: a systematic review and meta-analysis. Open Heart. 2019 Apr 9;6(1):e000922. doi: 10.1136/openhrt-2018-000922. eCollection 2019. PMID 31168371
- [Background] Otto CM, Nishimura RA, Bonow RO, Carabello BA, Erwin JP 3rd, Gentile F, Jneid H, Krieger EV, Mack M, McLeod C, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A, Toly C. 2020 ACC/AHA Guideline for the Management of Patients With Valvular Heart Disease: Executive Summary: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2021 Feb 2;143(5):e35-e71. doi: 10.1161/CIR.0000000000000932. Epub 2020 Dec 17. PMID 33332149
- [Background] Long L, Mordi IR, Bridges C, Sagar VA, Davies EJ, Coats AJ, Dalal H, Rees K, Singh SJ, Taylor RS. Exercise-based cardiac rehabilitation for adults with heart failure. Cochrane Database Syst Rev. 2019 Jan 29;1(1):CD003331. doi: 10.1002/14651858.CD003331.pub5. PMID 30695817
- [Background] Borg G. Borg's perceived exertion and pain scales. Leeds: Human Kinetics; 1998.
- [Background] Exercise tests in relation to cardiovascular function. Report of a WHO meeting. World Health Organ Tech Rep Ser. 1968;388:1-30. No abstract available. PMID 4968942
- [Background] Cider A, Carlsson S, Arvidsson C, Andersson B, Sunnerhagen KS. Reliability of clinical muscular endurance tests in patients with chronic heart failure. Eur J Cardiovasc Nurs. 2006 Jun;5(2):122-6. doi: 10.1016/j.ejcnurse.2005.10.001. Epub 2005 Oct 28. PMID 16257580
- [Background] Guralnik JM, Ferrucci L, Pieper CF, Leveille SG, Markides KS, Ostir GV, Studenski S, Berkman LF, Wallace RB. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci. 2000 Apr;55(4):M221-31. doi: 10.1093/gerona/55.4.m221. PMID 10811152
- [Background] Ekerstad N, Javadzadeh D, Alexander KP, Bergstrom O, Eurenius L, Fredrikson M, Gudnadottir G, Held C, Angerud KH, Jahjah R, Jernberg T, Mattsson E, Melander K, Mellbin L, Ohlsson M, Ravn-Fischer A, Svennberg L, Yndigegn T, Alfredsson J. Clinical Frailty Scale classes are independently associated with 6-month mortality for patients after acute myocardial infarction. Eur Heart J Acute Cardiovasc Care. 2022 Feb 8;11(2):89-98. doi: 10.1093/ehjacc/zuab114. PMID 34905049
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Orwelius L, Nilsson M, Nilsson E, Wenemark M, Walfridsson U, Lundstrom M, Taft C, Palaszewski B, Kristenson M. The Swedish RAND-36 Health Survey - reliability and responsiveness assessed in patient populations using Svensson's method for paired ordinal data. J Patient Rep Outcomes. 2017;2(1):4. doi: 10.1186/s41687-018-0030-0. Epub 2018 Feb 7. PMID 29757320
- [Background] Aadland E, Ylvisaker E. Reliability of the Actigraph GT3X+ Accelerometer in Adults under Free-Living Conditions. PLoS One. 2015 Aug 14;10(8):e0134606. doi: 10.1371/journal.pone.0134606. eCollection 2015. PMID 26274586
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- See also: .The National Board of Health and Welfare. National guidelines for cardiac disease. Stockholm 2015 [December 2017] — http://www.socialstyrelsen.se/kunskapsstod-och-regler/regler-och-riktlinjer/nationella-riktlinjer/riktlinjer-och-utvarderingar/hjartsjukvard/
- See also: Swedeheart annual report 2022 Uppsala Clinical Research Center. 2023. — http://www.ucr.uu.se/rikssvikt/om-rikssvikt/arsrapporter/arsrapporter/2022-arsrapport-swedeheart